CLINICAL TRIAL: NCT00327691
Title: The Effect Of LDL-Cholesterol, Lowering Beyond Currently Recommended Minimum Targets On Coronary Heart Disesse (CHD) Recurrence In Patients With Pre-Existing CHD
Brief Title: A Study to Determine the Degree of Additional Reduction in CV Risk in Lowering LDL Below Minimum Target Levels
Acronym: TNT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0981-117; A2581136
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Cardiovascular Disease; Cerebrovascular Accident; Coronary Heart Disease
Keywords: Major cardiovascular event; Major Coronary event; Revascularization
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Coronary Disease | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The primary objective of this study is to determine the degree of additional reduction in cardiovascular risk that was accrued to patients by lowering their LDL-C beyond the currently accepted minimum target level for patients with pre-existing CHD. Secondary objectives include the safety profile of this treatment strategy, its cost-effectiveness, effect on other atherosclerotic-related events and procedures, and total mortality.

ELIGIBILITY:
Inclusion Criteria:

Men and women age 35-75 who have evident CHD

Exclusion Criteria:

Known hypersensitivity to HMG CO-A reductase therapy, liver disease, evidence of secondary hyperlipidemia

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8600
Dates: Start 1998-04; Study Completion 2004-08

PRIMARY OUTCOMES:
The primary outcome is the time to occurrence of a major
cardiovascular event, defined as the composite outcome of the
following clinical endpoints
CHD death
Non-fatal/Non-procedure related MI
Resuscitated cardiac arrest or fatal/non-fatal stroke

SECONDARY OUTCOMES:
The occurrence of the following clinical events
Major coronary event (CHD death, non fatal myocardial infarction or resuscitated cardiac arrest)
any coronary event (major coronary event or CABG
PTCA, other revascularization procedure, procedure-related myocardial infarction, or documented angina)
cerebrovascular event (fatal or non fatal stroke, TIA)
peripheral vascular disease; hospitalization with primary diagnosis' of CHF
any cardiovascular event (any of the above); and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (246):
- United States (132):
  - Pfizer Investigational Site, Alabaster, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Hoover, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, Camp Pendleton, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Gainsville, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Inverness, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Tamarac, Florida
  - Pfizer Investigational Site, The Villages, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Canton, Georgia
  - Pfizer Investigational Site, Berwyn, Illinois
  - Pfizer Investigational Site, Blue Island, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Du Quoin, Illinois
  - Pfizer Investigational Site, Evanston, Illinois
  - Pfizer Investigational Site, Lake Forest, Illinois
  - Pfizer Investigational Site, Marion, Illinois
  - Pfizer Investigational Site, Pekin, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Beech Grove, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Scottsburg, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Lathe, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Edgewood, Kentucky
  - Pfizer Investigational Site, Erlanger, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bel Air, Maryland
  - Pfizer Investigational Site, Westminster, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Burlington, Massachusetts
  - Pfizer Investigational Site, Dearborn, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hill, Michigan
  - Pfizer Investigational Site, Sterling Heights, Michigan
  - Pfizer Investigational Site, West Bloomfield, Michigan
  - Pfizer Investigational Site, Duluth, Minnesota
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Maplewood, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Papillion, Nebraska
  - Pfizer Investigational Site, Manchester, New Hampshire
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Hawthorne, New York
  - Pfizer Investigational Site, Manlius, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Valhalla, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Eden, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Lorain, Ohio
  - Pfizer Investigational Site, Sandusky, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Lehighton, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Denton, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lackland Air Force Base, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (14):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Auchenflower, Queensland
  - Pfizer Investigational Site, Brisbane, Queensland
  - Pfizer Investigational Site, Chermside, Queensland
  - Pfizer Investigational Site, Greenslopes, Queensland
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Milton, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Hobart, Tasmania
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
  - Pfizer Investigational Site, Prahran, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Austria (3):
  - Pfizer Investigational Site, Feldkirch
  - Pfizer Investigational Site, Oberpullendorf
  - Pfizer Investigational Site, Vienna
- Belgium (7):
  - Pfizer Investigational Site, Aalst
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Godinne
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Lommel
  - Pfizer Investigational Site, Neerpelt
- Canada (18):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Nanaimo, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Greater Sudbury, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, St-foy, Quebec
- France (12):
  - Pfizer Investigational Site, Pessac, Cedex
  - Pfizer Investigational Site, Agen
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Roubaix
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Schwerte
  - Pfizer Investigational Site, Tostedt
  - Pfizer Investigational Site, Würzburg
- Ireland (2):
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Dublin
- Italy (6):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Cuneo
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Rome
  - Pfizer Investigational Site, Udine
- Netherlands (12):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Amersfoort
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Enschede
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Leiden
  - Pfizer Investigational Site, Nieuwegein
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Zwolle
- South Africa (5):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Sunninghill, Gauteng
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Parow
- Spain (9):
  - Pfizer Investigational Site, Córdoba, CORDOBA
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Donostia / San Sebastian
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Santiago de Compostela
  - Pfizer Investigational Site, Valladolid
  - Pfizer Investigational Site, Zaragoza
- Switzerland (5):
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Geneva
  - Pfizer Investigational Site, Lausanne
  - Pfizer Investigational Site, Lugano
  - Pfizer Investigational Site, Sankt Gallen
- United Kingdom (14):
  - Pfizer Investigational Site, Romford, ESSEX
  - Pfizer Investigational Site, London, GREATER LONDON
  - Pfizer Investigational Site, Aldershot, HAMPSHIRE
  - Pfizer Investigational Site, Farnborough, KENT
  - Pfizer Investigational Site, Blackpool, LANCASHIRE
  - Pfizer Investigational Site, Leicester, LEICESTERSHIRE
  - Pfizer Investigational Site, London, MIDDLESEX
  - Pfizer Investigational Site, Coventry, West Midlands
  - Pfizer Investigational Site, Coventry, WEST Midlands
  - Pfizer Investigational Site, Swindon, Wiltshire
  - Pfizer Investigational Site, Barnet
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Paisley
- Pfizer Investigational Site

REFERENCES:
- [Result] Waters DD, LaRosa JC, Barter P, Fruchart JC, Gotto AM Jr, Carter R, Breazna A, Kastelein JJ, Grundy SM. Effects of high-dose atorvastatin on cerebrovascular events in patients with stable coronary disease in the TNT (treating to new targets) study. J Am Coll Cardiol. 2006 Nov 7;48(9):1793-9. doi: 10.1016/j.jacc.2006.07.041. Epub 2006 Oct 17. PMID 17084252
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Vogt L, Bangalore S, Fayyad R, Melamed S, Hovingh GK, DeMicco DA, Waters DD. Atorvastatin Has a Dose-Dependent Beneficial Effect on Kidney Function and Associated Cardiovascular Outcomes: Post Hoc Analysis of 6 Double-Blind Randomized Controlled Trials. J Am Heart Assoc. 2019 May 7;8(9):e010827. doi: 10.1161/JAHA.118.010827. PMID 31020900
- [Derived] Bangalore S, Fayyad R, DeMicco DA, Colhoun HM, Waters DD. Body Weight Variability and Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004724. doi: 10.1161/CIRCOUTCOMES.118.004724. PMID 30571333
- [Derived] Kaasenbrood L, Ray KK, Boekholdt SM, Smulders YM, LaRosa JC, Kastelein JJP, van der Graaf Y, Dorresteijn JAN, Visseren FLJ. Estimated individual lifetime benefit from PCSK9 inhibition in statin-treated patients with coronary artery disease. Heart. 2018 Oct;104(20):1699-1705. doi: 10.1136/heartjnl-2017-312510. Epub 2018 Apr 5. PMID 29622600
- [Derived] Vallejo-Vaz AJ, Fayyad R, Boekholdt SM, Hovingh GK, Kastelein JJ, Melamed S, Barter P, Waters DD, Ray KK. Triglyceride-Rich Lipoprotein Cholesterol and Risk of Cardiovascular Events Among Patients Receiving Statin Therapy in the TNT Trial. Circulation. 2018 Aug 21;138(8):770-781. doi: 10.1161/CIRCULATIONAHA.117.032318. PMID 29618599
- [Derived] Ong KL, Waters DD, Fayyad R, Vogt L, Melamed S, DeMicco DA, Rye KA, Barter PJ. Relationship of High-Density Lipoprotein Cholesterol With Renal Function in Patients Treated With Atorvastatin. J Am Heart Assoc. 2018 Jan 22;7(2):e007387. doi: 10.1161/JAHA.117.007387. PMID 29358194
- [Derived] Ports WC, Fayyad R, DeMicco DA, Laskey R, Wolk R. Effectiveness of Lipid-Lowering Statin Therapy in Patients With and Without Psoriasis. Clin Drug Investig. 2017 Aug;37(8):775-785. doi: 10.1007/s40261-017-0533-0. PMID 28573499
- [Derived] Bangalore S, Fayyad R, Laskey R, DeMicco DA, Messerli FH, Waters DD. Body-Weight Fluctuations and Outcomes in Coronary Disease. N Engl J Med. 2017 Apr 6;376(14):1332-1340. doi: 10.1056/NEJMoa1606148. PMID 28379800
- [Derived] Stam-Slob MC, van der Graaf Y, Greving JP, Dorresteijn JA, Visseren FL. Cost-Effectiveness of Intensifying Lipid-Lowering Therapy With Statins Based on Individual Absolute Benefit in Coronary Artery Disease Patients. J Am Heart Assoc. 2017 Feb 18;6(2):e004648. doi: 10.1161/JAHA.116.004648. PMID 28214794
- [Derived] Deedwania PC, Pedersen TR, DeMicco DA, Breazna A, Betteridge DJ, Hitman GA, Durrington P, Neil A; TNT, CARDS and IDEAL Steering Committees and Investigators. Differing predictive relationships between baseline LDL-C, systolic blood pressure, and cardiovascular outcomes. Int J Cardiol. 2016 Nov 1;222:548-556. doi: 10.1016/j.ijcard.2016.07.201. Epub 2016 Jul 30. PMID 27513651
- [Derived] Byun YS, Lee JH, Arsenault BJ, Yang X, Bao W, DeMicco D, Laskey R, Witztum JL, Tsimikas S; TNT Trial Investigators. Relationship of oxidized phospholipids on apolipoprotein B-100 to cardiovascular outcomes in patients treated with intensive versus moderate atorvastatin therapy: the TNT trial. J Am Coll Cardiol. 2015 Apr 7;65(13):1286-1295. doi: 10.1016/j.jacc.2015.01.050. PMID 25835440
- [Derived] Arsenault BJ, Barter P, DeMicco DA, Bao W, Preston GM, LaRosa JC, Grundy SM, Deedwania P, Greten H, Wenger NK, Shepherd J, Waters DD, Kastelein JJ; Treating to New Targets (TNT) Investigators. Prediction of cardiovascular events in statin-treated stable coronary patients of the treating to new targets randomized controlled trial by lipid and non-lipid biomarkers. PLoS One. 2014 Dec 22;9(12):e114519. doi: 10.1371/journal.pone.0114519. eCollection 2014. PMID 25531109
- [Derived] Dorresteijn JA, Boekholdt SM, van der Graaf Y, Kastelein JJ, LaRosa JC, Pedersen TR, DeMicco DA, Ridker PM, Cook NR, Visseren FL. High-dose statin therapy in patients with stable coronary artery disease: treating the right patients based on individualized prediction of treatment effect. Circulation. 2013 Jun 25;127(25):2485-93. doi: 10.1161/CIRCULATIONAHA.112.000712. Epub 2013 May 14. PMID 23674398
- [Derived] Semb AG, Kvien TK, DeMicco DA, Fayyad R, Wun CC, LaRosa JC, Betteridge J, Pedersen TR, Holme I. Effect of intensive lipid-lowering therapy on cardiovascular outcome in patients with and those without inflammatory joint disease. Arthritis Rheum. 2012 Sep;64(9):2836-46. doi: 10.1002/art.34524. PMID 22576673
- [Derived] Huijgen R, Boekholdt SM, Arsenault BJ, Bao W, Davaine JM, Tabet F, Petrides F, Rye KA, DeMicco DA, Barter PJ, Kastelein JJ, Lambert G. Plasma PCSK9 levels and clinical outcomes in the TNT (Treating to New Targets) trial: a nested case-control study. J Am Coll Cardiol. 2012 May 15;59(20):1778-84. doi: 10.1016/j.jacc.2011.12.043. PMID 22575316 (Retraction: PMID 23729038 J Am Coll Cardiol. 2013 Apr 23;61(16):1751)
- [Derived] Mora S, Wenger NK, Demicco DA, Breazna A, Boekholdt SM, Arsenault BJ, Deedwania P, Kastelein JJ, Waters DD. Determinants of residual risk in secondary prevention patients treated with high- versus low-dose statin therapy: the Treating to New Targets (TNT) study. Circulation. 2012 Apr 24;125(16):1979-87. doi: 10.1161/CIRCULATIONAHA.111.088591. Epub 2012 Mar 29. PMID 22461416
- [Derived] Arsenault BJ, Boekholdt SM, Hovingh GK, Hyde CL, DeMicco DA, Chatterjee A, Barter P, Deedwania P, Waters DD, LaRosa JC, Pedersen TR, Kastelein JJ; TNT and IDEAL Investigators. The 719Arg variant of KIF6 and cardiovascular outcomes in statin-treated, stable coronary patients of the treating to new targets and incremental decrease in end points through aggressive lipid-lowering prospective studies. Circ Cardiovasc Genet. 2012 Feb 1;5(1):51-7. doi: 10.1161/CIRCGENETICS.111.960252. Epub 2011 Dec 1. PMID 22135385
- [Derived] Arsenault BJ, Barter P, DeMicco DA, Bao W, Preston GM, LaRosa JC, Grundy SM, Deedwania P, Greten H, Wenger NK, Shepherd J, Waters DD, Kastelein JJ; TNT Study Investigators. Prediction of cardiovascular events in statin-treated stable coronary patients by lipid and nonlipid biomarkers. J Am Coll Cardiol. 2011 Jan 4;57(1):63-9. doi: 10.1016/j.jacc.2010.06.052. PMID 21185503 (Retraction: PMID 23729037 J Am Coll Cardiol. 2013 Apr 23;61(16):1750)
- [Derived] Hyde CL, Macinnes A, Sanders FA, Thompson JF, Mazzarella RA, Faergeman O, van Wijk DF, Wood L, Lira M, Paciga SA. Genetic association of the CCR5 region with lipid levels in at-risk cardiovascular patients. Circ Cardiovasc Genet. 2010 Apr;3(2):162-8. doi: 10.1161/CIRCGENETICS.109.897793. Epub 2010 Feb 3. PMID 20130232
- [Derived] Waters DD. Clinical insights from the Treating to New Targets trial. Prog Cardiovasc Dis. 2009 May-Jun;51(6):487-502. doi: 10.1016/j.pcad.2009.01.001. PMID 19410683
- [Derived] Shepherd J, Kastelein JP, Bittner VA, Carmena R, Deedwania PC, Breazna A, Dobson S, Wilson DJ, Zuckerman AL, Wenger NK; Treating to New Targets Steering Committee and Investigators. Intensive lipid lowering with atorvastatin in patients with coronary artery disease, diabetes, and chronic kidney disease. Mayo Clin Proc. 2008 Aug;83(8):870-9. PMID 18674471
- [Derived] Shah SJ, Waters DD, Barter P, Kastelein JJ, Shepherd J, Wenger NK, DeMicco DA, Breazna A, LaRosa JC. Intensive lipid-lowering with atorvastatin for secondary prevention in patients after coronary artery bypass surgery. J Am Coll Cardiol. 2008 May 20;51(20):1938-43. doi: 10.1016/j.jacc.2007.12.054. PMID 18482661
- [Derived] Shepherd J, Kastelein JJ, Bittner V, Deedwania P, Breazna A, Dobson S, Wilson DJ, Zuckerman A, Wenger NK; TNT (Treating to New Targets) Investigators. Intensive lipid lowering with atorvastatin in patients with coronary heart disease and chronic kidney disease: the TNT (Treating to New Targets) study. J Am Coll Cardiol. 2008 Apr 15;51(15):1448-54. doi: 10.1016/j.jacc.2007.11.072. PMID 18402899
- [Derived] Barter P, Gotto AM, LaRosa JC, Maroni J, Szarek M, Grundy SM, Kastelein JJ, Bittner V, Fruchart JC; Treating to New Targets Investigators. HDL cholesterol, very low levels of LDL cholesterol, and cardiovascular events. N Engl J Med. 2007 Sep 27;357(13):1301-10. doi: 10.1056/NEJMoa064278. PMID 17898099
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0981-117&StudyName=The+study+is+to+determine+the+degree+of+additional+reduction+in+CV+risk+in+lowering+LDL+below+minimum+target+levels+